CLINICAL TRIAL: NCT02093403
Title: Phase I Study of Decitabine (Dacogen) and Selinexor (KPT-330) in Acute Myeloid Leukemia
Brief Title: Decitabine and Selinexor in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bhavana Bhatnagar (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Bhavana Bhatnagar, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-13182; NCI-2014-00559 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia; Adult Acute Myeloid Leukemia with T(8;21)(Q22;Q22); adult Acute Myeloid Leukemia with 11q23 (MLL) abnormalities; adult Acute Myeloid Leukemia with del(5q); adult Acute Myeloid Leukemia with inv(16)(p13;q22)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Decitabine; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (decitabine and selinexor) (Experimental): INDUCTION: Patients receive decitabine IV over 1 hour on days 1-10 and selinexor PO on days 11, 13, 18, 20, 25 and 27. Treatment repeats every 31 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive decitabine IV over 1 hour on days 1-5 and selinexor PO on days 6, 8, 13, 15, 20 and 22. Courses repeat every 31 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: decitabine; Drug: selinexor; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Drug: selinexor — Given PO
  Other Names: CRM1 nuclear export inhibitor KPT-330; KPT-330; selective inhibitor of nuclear export KPT-330; SINE KPT-330
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of Selinexor when given together with decitabine in treating patients with acute myeloid leukemia that has returned after treatment (relapsed) or does not respond to treatment (refractory). Drugs used in chemotherapy, such as decitabine and Selinexor, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of Selinexor (KPT-330) in combination with decitabine in patients with acute myeloid leukemia (AML).

II. To define the specific toxicities, maximum tolerated dose (MTD) and the dose limiting toxicity (DLT) of this combination.

III. To determine the Recommended Phase 2 Dose (RP2D) of this combination.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR). II. To determine the rate and duration of complete remission (CR) +/- hematological recovery of KPT-330 plus decitabine in AML.

III. To conduct pharmacodynamic studies by measuring the effect of this chemotherapy combination on the kinome, micronome and epigenome.

OUTLINE: This is a dose-escalation study of selinexor.

INDUCTION: Patients receive decitabine intravenously (IV) over 1 hour on days 1-10 and Selinexor orally (PO) on days 11, 13, 18, 20, 25 and 27. Treatment repeats every 31 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive decitabine IV over 1 hour on days 1-5 and Selinexor PO on days 6, 8, 13, 15, 20 and 22. Courses repeat every 31 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory AML
* Newly diagnosed elderly AML patients (> 60 years) unfit for intensive chemotherapy with cytarabine and anthracyclines are also eligible to this trial given that no clinically beneficial therapy exists for these patients
* Patients with secondary AML or therapy related disease (t-AML) are eligible; patients who received decitabine or 5-azacytidine as prior treatment for myelodysplastic syndrome (MDS) or AML remain eligible; however, none of these agents is permitted within 6 months of study entry
* If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Total bilirubin < 2.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
* Creatinine < 2.0 mg/d
* Glomerular filtration rate (GFR) > 50 mL/min
* New York Heart Association (NYHA) congestive heart failure (CHF) class II or better
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child]bearing potential; acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose
* Ability to understand and willingness to sign the written informed consent document
* Human immunodeficiency virus (HIV) infection without history of acquired immune deficiency syndrome (AIDS) and sufficiently high cluster of differentiation (CD)4 cells (> 400/mm^3) and low HIV viral loads (< 30,000 copies/ml plasma) not requiring anti-HIV therapy are eligible
* Patients must have recovered from the toxicity of prior therapy to less than grade 2

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients receiving any other investigational agents or patients that have received other investigational agents within 14 days of enrollment
* Patients with active central nervous system (CNS) malignancy; asymptomatic small lesions are not considered active; treated lesions may be considered inactive if they are stable for at least 3 months; patients with malignant cells in their cerebrospinal fluid (CSF) without CNS symptoms may be included
* Patients with history of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine that are not easily managed
* Major surgery within 2 weeks before day 1
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) ribonucleic acid (RNA) or HBsAg (hepatitis B virus [HBV] surface antigen)
* Patients with significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea
* History of seizures, movement disorders or cerebrovascular accident within the past 3 years prior to cycle 1 day 1
* Patients with macular degeneration, uncontrolled glaucoma, or markedly decreased visual acuity
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, myocardial infarction within 6 months prior to enrollment, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Pregnant women or women who are breastfeeding are excluded from this study; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patients with advanced malignant solid tumors are excluded
* Patients with renal failure (GFR < 50 mL/min) are excluded
* Patients that in the opinion of the investigators are significantly below their ideal body weight

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-11-26 (Actual); Study Completion 2016-11-26 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose where at most one patient experiences DLT with the next higher dose having at least 2 patients who experience DLT graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 31 days
Incidence of severe (grade 3+) adverse events or toxicities assessed by NCI CTCAE version 4.03 | Up to 3 years
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Tolerability of the regimen defined by the number of patients who required dose modifications and/or dose delays | Up to 3 years
Proportion of patients who go off treatment due to adverse reactions | Up to 3 years

SECONDARY OUTCOMES:
Overall response rate | Up to 3 years
  Responses will be summarized by simple descriptive summary statistics across all dose levels. Overall response rate will estimated at the MTD and defined as the number of patients who achieve any level of clinical response (e.g. CR, incomplete blood count recovery, morphologic CR) divided by the total number of evaluable patients (i.e. any patient who received at least one dose of study treatment).
Complete response rate | Up to 3 years
  Responses will be summarized by simple descriptive summary statistics across all dose levels. Complete response rate will be estimated in those patients treated at the MTD.
Change in expression of XPO1 | Baseline to up to day 31 of course 1
  Changes in expression of these markers across time will be explored by dose level graphically. Relationships between baseline expression levels and changes in expression levels with response and certain toxicities will also be explored graphically (e.g. side-by-side boxplots) and with quantitative summaries. Confidence intervals will be presented as the primary method of analysis. Correlations among expression of the genes, micro-ribonucleic acids (miRs), and methylated signatures will be evaluated using scatterplots and the Spearman-rank correlation coefficient.
Change in expression of genes associated with XPO1 | Baseline to up to day 31 of course 1
  Changes in expression of these markers across time will be explored by dose level graphically. Relationships between baseline expression levels and changes in expression levels with response and certain toxicities will also be explored graphically (e.g. side-by-side boxplots) and with quantitative summaries. Confidence intervals will be presented as the primary method of analysis. Correlations among expression of the genes, miRs, and methylated signatures will be evaluated using scatterplots and the Spearman-rank correlation coefficient.
Change in expression of miRs associated with XPO1 | Baseline to up to day 31 of course 1
  Changes in expression of these markers across time will be explored by dose level graphically. Relationships between baseline expression levels and changes in expression levels with response and certain toxicities will also be explored graphically (e.g. side-by-side boxplots) and with quantitative summaries. Confidence intervals will be presented as the primary method of analysis. Correlations among expression of the genes, miRs, and methylated signatures will be evaluated using scatterplots and the Spearman-rank correlation coefficient.
Change in expression of methylated signatures | Baseline to up to day 31 of course 1
  Changes in expression of these markers across time will be explored by dose level graphically. Relationships between baseline expression levels and changes in expression levels with response and certain toxicities will also be explored graphically (e.g. side-by-side boxplots) and with quantitative summaries. Confidence intervals will be presented as the primary method of analysis. Correlations among expression of the genes, miRs, and methylated signatures will be evaluated using scatterplots and the Spearman-rank correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Bhatnagar, DO, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Bhatnagar B, Zhao Q, Mims AS, Vasu S, Behbehani GK, Larkin K, Blachly JS, Blum W, Klisovic RB, Ruppert AS, Orwick S, Oakes C, Ranganathan P, Byrd JC, Walker AR, Garzon R. Selinexor in combination with decitabine in patients with acute myeloid leukemia: results from a phase 1 study. Leuk Lymphoma. 2020 Feb;61(2):387-396. doi: 10.1080/10428194.2019.1665664. Epub 2019 Sep 23. PMID 31545113
- See also: The Jamesline — http://cancer.osu.edu